CLINICAL TRIAL: NCT05205681
Title: The Role of Imaging in the Diagnosis of Acute Appendicitis During the COVID-19 Pandemic: a Retrospective Cohort Study
Brief Title: The Role of Imaging in the Diagnosis of Acute Appendicitis During the COVID-19 Pandemic
Status: Completed | Type: Observational
Sponsor: University College London Hospitals (Other)
Responsible Party: Principal Investigator, Dr Gerardo Perrotta, Trust Grade Doctor in General Surgery, University College London Hospitals
Other Study IDs: NARCO2021
Record Dates: First submitted 2022-01-07; First posted 2022-01-25 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Appendicitis
Keywords: appendicitis; COVID-19; negative appendicectomy rate; computer tomography; ultrasonography; pre-operative imaging
MeSH Terms: conditions — Appendicitis; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pandemic Group: All patients who underwent emergency appendicectomy for suspected acute appendicitis between March 2020 and February 2021
  Interventions: Diagnostic Test: Pre-operative imaging
- Control Group: All patients who underwent emergency appendicectomy for suspected acute appendicitis between March 2019 and February 2020
  Interventions: Diagnostic Test: Pre-operative imaging

INTERVENTIONS:
Diagnostic Test: Pre-operative imaging — Use of pre-operative imaging or the diagnosis of acute appendicitis

SUMMARY:
This is a retrospective observational study in the form of a cohort study evaluating the use of pre-operative imaging for the diagnosis of acute appendicitis in a tertiary centre during the first and second waves of the COVID-19 pandemic in the United Kingdom. The study group includes all patients who underwent emergency appendicectomy for suspected acute appendicitis between March 2020 and February 2021, while the control group includes all patients who underwent emergency appendicectomy for suspected acute appendicitis between March 2019 and February 2020. The final histology will be used as primary outcome, as the study hypothesis is that increasing the use of pre-operative imaging will reduce the negative appendicectomy rate.

ELIGIBILITY:
Inclusion Criteria:

* Patients of all ages who underwent emergency appendicectomy (either laparoscopic or open) for suspected acute appendicitis
* Patients of all ages who underwent partial ileo-caecectomy or right hemicolectomy for suspected acute appendicitis

Exclusion Criteria:

* Patients who underwent elective interval appendicectomy for a previous appendiceal phlegmon
* Patients who underwent appendicectomy or right hemicolectomy for appendiceal tumours
* Patients who underwent diagnostic laparoscopy for suspected acute appendicitis, where the appendix was not removed

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive patients operated at a tertiary centre
Sampling Method: Non-Probability Sample
Enrollment: 313 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Negative Appendicectomy Rate (NAR) | Up to 3 weeks post-operatively (when final Histology is ready)
  Number of patients with final histology negative for acute appendicitis

SECONDARY OUTCOMES:
Post-Operative Length of Stay | Assessed on day 30 after the completion of the study
  Post-operative length of hospital stay (from post-operative day 1)
Post-Operative Complications Rate | Within 30 post-operative days
  Number of patients who had post-operative complications

CONTACTS AND LOCATIONS:
Overall Officials: Gerardo Perrotta, MD, Principal Investigator — University College London Hospitals
Locations (1):
- University College London Hospitals NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Perrotta G, Geropoulos G, Bhan C. The role of imaging in the diagnosis of acute appendicitis during the COVID-19 pandemic: a retrospective cohort study. Updates Surg. 2023 Jan;75(1):205-208. doi: 10.1007/s13304-022-01426-y. Epub 2022 Nov 24. PMID 36422811